CLINICAL TRIAL: NCT04877197
Title: Behavioral Activation Delivered Via Home-based Telehealth to Improve Functioning in Cardiovascular Disease Patients Recently Discharged From Inpatient Care
Acronym: VA HEART
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: F3377-R; RX003377-01A2 (Other Grant/Funding Number: VA Rehabilitation Research and Development Service)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Depression; Cardiovascular Diseases
Keywords: Veterans; Mental Health; Veterans Health; Cardiovascular Diseases
MeSH Terms: conditions — Depression; Cardiovascular Diseases; Psychological Well-Being | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The investigators will use a 2x4 (treatment by time) repeated measures RCT crossover design (baseline, post-treatment, 3 & 9-month follow-up; crossover for standard treatment group at 9 months). At the 9 month point, the comparison group will have the option of receiving the intervention.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The only members of the research team who will be aware of randomization assignment will be the project therapists, the research coordinator, and the statistical analyst in charge of randomization. The outcomes assessor and investigator will be blinded to subject assignment, and though treating physicians will be informed of their patient's participation in the study, they will be blinded to treatment condition. Patients will be given instructions not to disclose their treatment assignment to their treating physicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BA-HT (Experimental): Behavioral Activation for depression delivered via home-based telehealth (BA-HT) will be implemented over 12, weekly 50-minute sessions via VA approved telehealth software.
  Interventions: Behavioral: BA-HT
- Standard Care (Active Comparator): Best practices standard care delivery for post-CVD hospitalization as regularly implemented at the RHJ VAMC. Standard care may include all or some of the following: post-operative follow up, referral to VA primary care clinic at 1 month post-procedure, primary care visit with VA mandated assessments of pain and depression with referral for these conditions, referral to facility-based or home-based cardiac rehabilitation program as appropriate. All participants in this condition will be referred to mental health care. In addition, these participants will receive a weekly telephone call from project staff during which time supportive questioning about patient progress and general mood and recovery.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: BA-HT — Behavioral Activation for depression delivered via home-based telehealth (BA-HT) will be implemented over 12, weekly 50-minute sessions via VA approved telehealth software.
  Other Names: Behavioral Activation for depression delivered via home-based telehealth
  Arms: BA-HT
Other: Standard Care — Best practices standard care delivery for post-CVD hospitalization as regularly implemented at the RHJ VAMC. Standard care may include all or some of the following: post-operative follow up, referral to VA primary care clinic at 1 month post-procedure, primary care visit with VA mandated assessments of pain and depression with referral for these conditions, referral to facility-based or home-based cardiac rehabilitation program as appropriate. All participants in this condition will be referred to mental health care. In addition, these participants will receive a weekly telephone call from project staff during which time supportive questioning about patient progress and general mood and recovery.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to demonstrate whether Behavioral Activation for depression delivered via home based telehealth (BA-HT) is effective in improving social and role functioning in Veterans recently discharged from Cardiovascular disease (CVD-related) inpatient care. Eligible participants will receive either (1) twelve sessions of BA-HT or (2) standard best practices post CVD hospitalization care.

Study participants will be 132 Veterans discharged from the Ralph H. Johnson VA Medical Center inpatient care facilities with CVD diagnoses corresponding to ICD 10 codes I20-I25 (120 unstable angina, stable angina; 121 NSTEMI, STEMI, initial encounter; 122 NSTEMI, STEMI, subsequent encounter; 124 acute coronary syndrome; 125 coronary arteriosclerosis with angina). They will be male or female, age 21 and above, and with approximately 40-50% minority representation. There will be assessment at baseline, 1 week post treatment, as well as 3 and 9-months post treatment.

The investigators predict that BA-HT will more effectively increase social role and activity functioning, activity, mood and reduce 9-month re-hospitalization compared to current best-practices post-discharge care among patients scoring at least moderately depressed on the PROMIS Depression scale one week following hospital discharge for a CVD event.

DETAILED DESCRIPTION:
Following hospital discharge, risk of depression is significantly increased in cardio-vascular disease (CVD) patients. Moreover, CVD patients with depression face reduced functioning, increased morbidity and mortality, and diminished quality of life. Unfortunately, most depressed CVD patients do not receive appropriate evidence-based care for their depression, often because they are unable to, or fearful of travelling to providers for the regimen of 8-12 weekly visits of evidence-based psychotherapy such as Behavioral Activation (BA). The group developed, evaluated and subsequently implemented in VA clinics, the first VA program to use home based telehealth to deliver BA for depression to elderly Veterans. The investigators now propose to evaluate the ability of this evidence based treatment and delivery model (BA for depression via home-telehealth) to reduce functional impairment and improve recovery in depressed Veterans who have experienced a CVD event-related hospitalization.

The specific aims of this project are:

1. To compare effectiveness of Behavioral Activation for depression delivered via Home-based Telehealth- to standard post-CVD hospital discharge best-practices care in a 2x4 (treatment by time) repeated measures RCT crossover design (baseline, post-treatment, 3 & 9-month follow-up; crossover for standard treatment group at 9 months) with 132 CVD Veteran patients evincing depression in terms of central outcomes of functioning (PROMIS Functioning and Global Health scales) and emotional symptoms (PROMIS Depression and Anxiety scales) and secondary objective outcomes related to activity (actigraphy data). At the 9 month point, the comparison group will have the option of receiving the intervention (thus complementing the RCT with a crossover phase).
2. To repeat these comparisons with sex and age as independent variables.
3. To evaluate BA-HT with respect to its effects on exploratory outcomes, including re-hospitalization.

The investigators predict that evidence-based psychotherapy for depression (i.e., Behavioral Activation) delivered via home based telehealth will more effectively increase social role and activity functioning, activity, mood and reduce 6-month re-hospitalization (exploratory hypothesis), compared to current best-practices post-discharge care among patients scoring at least moderately depressed on the PROMIS Depression scale one week following hospital discharge for a CVD event.

If effective, this innovative treatment and delivery strategy will enhance global functioning, improve quality of life, and reduce costs to Veterans and the VA. Importantly, the proposed strategy leverages existing VA infrastructure and capabilities so that BA-HT could be immediately offered throughout VA as a preventative measure to enhance resiliency.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced one of the ICD 10 I20-I25 CVD events:

  * 120 unstable angina
  * stable angina
  * 121 NSTEMI
  * STEMI
  * initial encounter
  * 122 NSTEMI
  * STEMI
  * subsequent encounter
  * 124 acute coronary syndrome
  * 125 coronary arteriosclerosis with angina and/or
  * Valve repair, valve replacement, Transcatheter Aortic Valve Implantation (TAVI/TAVR), Pacemaker Implantation in the past 6 months, Implantable Cardioverter Defibrillators (ICDs) in the past 6 months; Left Ventricular Assist Device in the past 6 months; Ablation Therapy; Watchman Implant; and
* Discharged from the RHJ VAMC inpatient care facilities
* Diagnosis of Major Depressive Disorder on the basis of the Structured Clinical Interview for DSM 5 (First, Williams, Karg, & Spitzer, 2015)

Exclusion Criteria:

* Coronary Artery Bypass Grafting (CABG)
* Having a household member who is already enrolled in the study
* Active psychosis or significant dementia at screening
* Suicidal ideation with clear intent
* Current alcohol use disorder rated severe
* Concurrent enrollment in another clinical trial for depression

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PROMIS Ability to Participate in Social Roles and Activities | 13 weeks
  This measure of functioning assesses one's perceived ability to perform usual social roles and activities. Items are worded negatively in terms of perceived limitations and are reverse-coded with higher scores represent fewer limitations. Each of the 8 items are scored 1 to 5 and totaled raw scores are used to derive T-scores, scaled to US general population estimates. In addition to PROMIS general validation efforts, evidence for reliability, construct validity, and sensitivity to change with cardiovascular surgery patients was provided by Flynn et al. (2015).
PROMIS Satisfaction with Participation in Social Roles | 13 weeks
  This 8-item measure (items rated 1 to 5, higher scores corresponding to higher satisfaction), assesses satisfaction related to one's ability and performance of work, routine activities, and family activities and is responsive to change over time (Hahn et al., 2016). Thus, this measure complements purely functional assessment of capabilities with assessment of participant's impression of the quality their functioning.
PROMIS Physical Function with Mobility Aid | 13 weeks
  This 11-item measure (high scores correspond to better mobility) is rated 1 to 5 (unable to do to "without any difficulty") and assesses self-report regarding many basic physical aspects of Activities of Daily Living. Both upper and lower extremity functioning is assessed, as well as instrumental activities.

CONTACTS AND LOCATIONS:
Overall Officials: Ron E. Acierno, PhD MS BA, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No